CLINICAL TRIAL: NCT06642116
Title: Evaluation of the Safety and Performance of a Bioresorbable Nasal Dressing Containing Mometasone Furoate
Acronym: ENHANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-4
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Rhinosinusitis Chronic; Wound Healing; Sinus Surgery; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OCEAN (Experimental): Application of OCEAN after nasal/sinus surgery
  Interventions: Device: OCEAN

INTERVENTIONS:
Device: OCEAN — Biodegradable nasal dressing

SUMMARY:
The objective of this study is to investigate the safety and performance of OCEAN® as an adjunct in wound healing after nasal/sinus surgery by using OCEAN® in patients undergoing nasal/sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older
2. Patient is scheduled to undergo bilateral endoscopic sinus surgery for Chronic Rhinosinusitis with nasal polyps (CRSwNP) or Chronic Rhinosinusitis without nasal polyps (CRSsNP)
3. Patient is willing and able to comply with all study elements as indicated by their written informed consent
4. Patients with a pre-operative Lund-MacKay score of ≥ 6.

Exclusion Criteria:

1. Patient is pregnant or nursing
2. Patients with a history of chronic epistaxis or experienced a significant epistaxis event (defined as epistaxis requiring medical intervention) in the past 3 months
3. Patients with a platelet disorder
4. Patients with a known or suspected allergy to device components
5. Patients with known hemophilia
6. Patients with insulin dependent diabetics
7. Patients with an oral steroid dependent condition
8. Patients with glaucoma, ocular hypertension, posterior subcapsular cataracts
9. Patients with a (previous) diagnosis of Samter's Triad (aspirin-exacerbated respiratory disease (AERD))
10. Patients that require nasal ointments or creams at time of device placement
11. Patients with a neurological, medical, psychiatric condition, or social circumstance that would potentially increase risk, interfere with study participation, or confound interpretation of study data
12. Patients with plans to (or otherwise anticipate the need to) undergo an ear, nose, throat (ENT) procedure within the 90 day study follow up
13. Patients participating in another clinical research study (within 30 days prior to screening up till 90 days post-operative).
14. Patients that used any form of corticosteroid or immunologics within 2 weeks prior to sinus surgery or during follow-up to day 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to 25 days after surgery
  Rate of serious adverse events related to the use of the OCEAN bioresorbable nasal dressing post nasal surgery
Performance | Up to 25 days after surgery
  Endoscopic evaluation of aspects of wound healing as assessed using the Lund-Kennedy Endoscopic Score System (LKS).
  The LKS assesses various factors like edema, crusting, discharge, polyps, and mucosal inflammation. Each parameter is scored from 0 to 2, with 0 being normal and 2 representing severe findings. Higher scores on the Lund-Kennedy Scale indicate a worse outcome, reflecting more severe disease or poor wound healing.
  Minimum Value: 0 (This represents no signs of inflammation or disease); Maximum Value: 20 (This indicates the most severe signs of disease or inflammation)